CLINICAL TRIAL: NCT06059651
Title: The Effects of Metabolic & Bariatric Surgery on Lipid Metabolism, Myeloid-Derived Suppressor Cells, and Cancer Cell Biology
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Justin Brown, Director, Cancer Metabolism Program, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-026
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Metabolic Networks and Pathways; Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Cohort #1 (within-subject) will enroll up to 10 women with class III obesity who plan to undergo Roux-en-Y metabolic and bariatric surgery as a standard of obesity care. Subjects will complete study measures preoperatively and one year postoperatively.
  Interventions: Procedure: Metabolic & Bariatric Surgery
- Cohort 2: Cohort #2 (between-subject) will enroll up to 10 women with a history of class III obesity who underwent Roux-en-Y metabolic and bariatric surgery as a standard of obesity care approximately one year before enrollment. Subjects in this cohort will be matched on demographic and clinical variables to those in Cohort #1.
  Interventions: Procedure: Metabolic & Bariatric Surgery

INTERVENTIONS:
Procedure: Metabolic & Bariatric Surgery — Roux-en-Y metabolic and bariatric surgery

SUMMARY:
This study aims to determine the relationship between lipid kinetics changes and blood immunosuppressive cells by metabolic surgery in two patient cohorts.

ELIGIBILITY:
For an eligible subject, all the following must be answered "yes":

* Biological female sex
* Age >=35 and <=60 years (including pre- and postmenopausal)
* Self-reported white or black race
* The study will enroll approximately 50% white and 50% black subjects
* Body mass index >/=40 kg/m2
* Have a diagnosis of hyperlipidemia (high triglycerides and LDL-cholesterol) or in treatment with any medication for hyperlipidemia at enrollment
* Ability to provide written informed consent
* Allow the collection and storage of biospecimens and data for future use
* Not having yet started the pre-op liquid diet before the bariatric surgery

For an eligible subject, all the following must be answered "no":

* Have type one or type two diabetes
* Use of anti-inflammatory medications, such as glucocorticoids or non-steroidal anti-inflammatory medications, within the past 15 days
* Use of medication approved for obesity management, including, but not limited to, phentermine-topiramate (Qsymia), orlistat (Xenical), naltrexone-bupropion (Contrave), liraglutide (Saxenda), and semaglutide (Wegovy)
* History of cancer of any type
* History of chronic conditions known to cause inflammation, such as tuberculosis, autoimmune disease, and human immunodeficiency virus
* An acute history (within the past 60 days) or confirmed or suspected SARS-CoV-2 (COVID-19) infection
* Currently pregnant, breastfeeding, or planning to become pregnant within the next 52 weeks
* Currently participating in another study with competing outcomes
* Any other situation that, in the opinion of the investigator, would negatively impact subject safety or successful compliance with the protocol

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The study population will include women with class III obesity who plan to undergo or have completed treatment with metabolic and bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in insulin-inhibited adipose tissue lipolysis | Baseline, week 52
Change in the number of circulating myeloid-derived suppressor cells | Baseline, week 52

CONTACTS AND LOCATIONS:
Overall Officials: Justin Brown, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Resarch Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No